CLINICAL TRIAL: NCT04586543
Title: A Clinical Trial of Selegiline Plus Docetaxel for the Treatment of Metastatic, Castrate-resistant Prostate Adenocarcinoma
Brief Title: Clinical Trial of Selegiline Plus Docetaxel for the Treatment of Metastatic, Castrate-resistant Prostate Adenocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: László Mangel (Other)
Collaborators: E-Group ICT Software Informatikai Zrt. (Unknown)
Responsible Party: Sponsor-Investigator, László Mangel, Prof MD, University of Pecs
Organization: University of Pecs (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAO201901; 2019-002685-12 (EudraCT Number)
Record Dates: First submitted 2020-09-30; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Metastatic Castration-resistant Prostate Cancer; Adenocarcinoma of the Prostate
Keywords: selegiline; hormone-refractory prostate cancer
MeSH Terms: interventions — Selegiline; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selegiline+ Docetaxel (Experimental): Selegiline and plus Docetaxel
  Interventions: Drug: Selegiline; Drug: Docetaxel
- Docetaxel (Active Comparator): Docetaxel
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Selegiline — 10 mg selegiline tablet per day
  Arms: Selegiline+ Docetaxel
Drug: Docetaxel — 75mg/m2 docetaxel infusion every 3 weeks for maximum of 12 cycles

SUMMARY:
The objective of this clinical study is to evaluate the effectiveness and safety of selegiline plus docetaxel therapy compared to the standard of care - docetaxel therapy - among patients diagnosed with metastatic, castrate-resistant prostate adenocarcinoma.

DETAILED DESCRIPTION:
Prostate cancer is one of the leading cause of cancer death among males worldwide. The objective of this phase II, randomized, controlled, open label study is to evaluate the effectiveness and safety of MAO-B (Monoamine oxidases-B) inhibitor selegiline plus docetaxel therapy. Patients diagnosed with metastatic, castrate-resistant prostate adenocarcinoma are randomly divided into two groups. One group (control arm) receives docetaxel (75 mg/m2 IV every 3 weeks for maximum of 12 cycles). Another group (experimental arm) receives docetaxel (75 mg/m2 IV every 3 weeks for maximum of 12 cycles) plus selegiline (daily 10 mg tablet). Patients are followed up for 36 months or until the end of the trial, death or withdraw from this study due to other reasons. The primary endpoint of this study is the proportion of patients without progression at month 9. The secondary endpoint is proportion of patients without progression at month 12/18, progression-free survival, overall survival, duration of PSA response, radiological response rate, PSA response rate, health-related quality of life and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older male patients,
2. Histologically or cytologically confirmed prostate adenocarcinoma
3. Radiologically confirmed metastatic disease,
4. Eligibility to receive oral therapy,
5. Suitable for docetaxel therapy,
6. Patients with castration-resistant prostate carcinoma who eligible to first-line docetaxel therapy or patients with castration-resistant prostate cancer who progressed after second-generation hormone therapy (abiraterone or enzalutamide) with pre-chemotherapy indication and eligible to second-line docetaxel therapy
7. At least 4 weeks has elapsed between the last antiandrogenic therapy and the inclusion (at least 6 weeks in case of bicalutamide),
8. Planned docetaxel treatment,
9. Eastern Cooperative Oncology Group (ECOG) performance status: ≤ 2,
10. Estimated life expectancy of more than 12 weeks,
11. Adequate analgesic therapy as required;
12. Patients must be able to follow the diet and medical instructions,
13. Use of effective contraception in men of childbearing age,
14. Provision of signed, written information consent

Exclusion Criteria:

1. De novo metastatic patients who needs immediate docetaxel therapy;
2. Within 4 weeks prior to randomisation, the patient has received other study medication or failed to recover from any adverse events caused from a previously administered study drug
3. ≥ Grade 2 anticancer therapy-related toxicity (except alopecia),
4. Has had radiotherapy or immunotherapy within 4 weeks prior to treatment,
5. Has had a surgery within 4 weeks prior to treatment,
6. Known or suspected brain metastasis (stable patients with locally treated, asymptomatic brain metastases are not excluded),
7. Inadequate laboratory function:

   1. Absolute neutrophil count <1.5 x 109 /L (1,500 per mm3),
   2. Platelet count < 100 x 109 /L (100 000 per mm3),
   3. Hemoglobin ≤9.0 g/dL,
   4. Serum bilirubin > ULN,
   5. AST or ALT

   i.>2.5 x ULN in patient without liver metastases, ii.>5x ULN in patients with liver metastases.
8. Cardiological status:

   1. Uncontrolled hypertension (BP ≥ 150/95 with hypertension treatment)
   2. Heart failure (NYHA III or higher),
   3. Current or former diagnosis of cardiomyopathy,
   4. LVEF ≤ 50%,
   5. Atrial fibrillation with >100bpm pulse,
   6. Unstable ischemic heart disease (myocardial infarction within 6 months or angina that require more than one nitrate therapy each week).
9. Other uncontrolled or severe systemic disease, active infection, hepatitis B, hepatitis C, HIV,
10. Uncontrolled seizure disorder,
11. Active gastric and duodenal ulcers,
12. Recurrent nausea and vomiting, chronic gastrointestinal disease or intestinal resection that prevents proper absorption,
13. Severe psychiatric illness (including but not limited to manic psychiatric disorder, schizophrenia, bipolar disorder, major depression requiring hospitalization) or social disturbance that limits eligibility for examination,
14. History of other malignancy within the last 5 years (except properly treated basalioma or squamous cell carcinoma of the skin and in situ carcinoma),
15. History of allergic reaction to phenelzine, selegiline or other monoamine oxidase inhibitors (MAOIs) biological agents or similar chemical ingredients,
16. History of allergic reaction to docetaxel therapy or its ingredients,
17. Significant peripheral neuropathy (≥ Grade 2),
18. Selegiline is contra-indicated for concomitant use with:

    1. Certain narcotic analgesics (eg. pethidine),
    2. Drugs that enhance the sympathetic nervous system,
    3. Other MAO inhibitors,
    4. Drugs similar to MAO inhibitors,
    5. Selective serotonin reuptake inhibitors (SSRIs) or serotonin norepinephrine reuptake inhibitors (SNRIs),
    6. Tricyclic antidepressants.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 110 (Estimated)
Dates: Start 2020-05-18 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients without progression at month 9 | 12 months
  Proportion of patients without progression at month 9. Progression can be identified by clinical symptoms, PSA levels, or radiographic imaging as follows, based on PCWG2 criteria:
  1. Progression based on clinical symptoms:
     1. Decline in ECOG performance status (≥ grade 3),
     2. Initiation of newly adjusted chronic opioid analgesic therapy, which may be,
     i.Use of oral opioid for at least 3 weeks ii.Use of parenteral opioid for at least 7 days c.Necessity to initiate alternative cytotoxic chemotherapy or other active systemic oncology treatment d.Immediate need for radiation or surgical intervention to treat tumor progression OR
  2. PSA progression: Date at which the PSA level is increased by at least 25% relative to nadir and at least 2 ng / mL absolute increase compared to the nadir. Values are confirmed 4-6 weeks later by a test.
     OR
  3. Radiological
     1. Progression by RECIST 1.1.
     2. Bone scan progression: A total of ≥ 2 new lesion compared to baseline

SECONDARY OUTCOMES:
Proportion of patients without progression at month 12 | 15 months
Proportion of patients without progression at month 18 | 21 months
Progression-free survival (biochemical, clinical, radiological | 5 years
Overall survival | 5 years
Duration of PSA response | 5 years
Radiological Response Rate | 5 years
PSA Response Rate | 5 years
Health-Related Quality of Life | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pécs, Clinical Centre, Department of Oncotherapy, Pécs, Baranya, Hungary